CLINICAL TRIAL: NCT06135974
Title: Phase 1 Trial of Multi-strain Lactobacillus Crispatus Vaginal Live Biotherapeutic Product
Brief Title: Vaginal lIve Biotherapeutic RANdomized Trial
Acronym: VIBRANT
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Ragon Institute of MGH, MIT and Harvard (Other); Centre for the AIDS Programme of Research in South Africa (Network)
Responsible Party: Principal Investigator, Caroline Mitchell, Associate Professor of Obstetrics, Gynecology & Reproductive Biology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VMRC001
Record Dates: First submitted 2023-11-02; First posted 2023-11-18 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Bacterial Vaginosis
Keywords: live biotherapeutic; bacterial vaginosis; vaginitis
MeSH Terms: conditions — Vaginosis, Bacterial; Vaginitis | interventions — Metronidazole

STUDY DESIGN:
Intervention Model Description: This is a randomized trial with 5 arms
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study product is labeled in a blinded manner with a code. Only pharmacy will have the link to the code and treatment assignment. However, the one arm starting study product during antibiotic treatment will be unblinded for both participants and investigators. However, the laboratory staff conducting the analyses for the primary and secondary outcomes will remain masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Placebo (Placebo Comparator): Vaginal placebo tablet administered daily for 7 days starting after antibiotic treatment
  Interventions: Drug: Placebo; Drug: Metronidazole Oral
- LC106 7 days (Experimental): Vaginal live biotherapeutic product with 6 strains of L. crispatus, administered daily for 7 days after antibiotic treatment
  Interventions: Drug: LC106; Drug: Metronidazole Oral
- LC106 3 days (Experimental): Vaginal live biotherapeutic product with 6 strains of L. crispatus, administered daily for 3 days after antibiotic treatment and packaged with 4 tablets of placebo to maintain masking (so a total of 7 tablets)
  Interventions: Drug: LC106; Drug: Metronidazole Oral
- LC106 7 days, early start (Experimental): Vaginal live biotherapeutic product with 6 strains of L. crispatus, administered daily for 7 days starting on the 3rd day of antibiotic treatment
  Interventions: Drug: LC106; Drug: Metronidazole Oral
- LC115 (Experimental): Vaginal live biotherapeutic product with 15 strains of L. crispatus, administered daily for 7 days after antibiotic treatment
  Interventions: Drug: LC115; Drug: Metronidazole Oral

INTERVENTIONS:
Drug: LC106 — Tablet containing at least 2 x 10^6 CFU/tablet, and comprised of 6 strains of Lactobacillus crispatus
  Arms: LC106 3 days; LC106 7 days; LC106 7 days, early start
Drug: LC115 — Tablet containing at least 2 x 10^6 CFU/tablet, and comprised of 15 strains of Lactobacillus crispatus
  Arms: LC115
Drug: Placebo — Vaginal tablets containing primarily microcrystalline cellulose and no live bacteria
  Arms: Placebo
Drug: Metronidazole Oral — Metronidazole tablet orally twice daily for 7 days

SUMMARY:
The goal of this randomized clinical trial is to evaluate safety and biologic effect of a multi-strain vaginal L. crispatus live biotherapeutic product (LBP) in people receiving antibiotic treatment for bacterial vaginosis (BV). The main question[s] it aims to answer are whether the intervention is safe, and whether the strains of L. crispatus will colonize recipients' vagina. The study will evaluate one LBP with 6 strains of L. crispatus (LC106) and one LBP with 15 strains (LC115) vs. placebo.

Participants will:

* be treated with oral antibiotics for BV
* receive 7 days of vaginal study product
* collect daily home swabs and make short daily diary entries for 5 weeks, including the week of antibiotic treatment and the week of study product treatment.

Researchers will compare the 3 groups receiving different dosing strategies of LC106 and 1 group receiving LC115 vs. 1 group receiving placebo to see if the live biotherapeutic strains colonize the vagina after antibiotic treatment for BV.

DETAILED DESCRIPTION:
This is a Phase I randomized trial of a novel live biotherapeutic intervention containing multiple strains of L. crispatus.

L. crispatus is a species of Lactobacillus commonly found in the human vagina, which is associated with optimal reproductive health outcomes. Detection of, and dominance of the community by, L. crispatus is associated with lower risk for bacterial vaginosis (BV), but no intervention to date has demonstrated the ability to durably shift the vaginal microbiome to L. crispatus dominance in a majority of treated people.

In this study, we will compare safety and biologic effects of two formulations of a consortia of L. crispatus strains, and a variety of dosing strategies in women with BV who receive antibiotic treatment. Our primary outcome is colonization with any of the L. crispatus strains contained in the live biotherapeutic product. All participants will have menses suppressed with either injectable progesterone contraception or continuous oral contraceptive pills for the duration of the study.

All participants will receive 7 days of oral metronidazole (500mg twice daily) and will be randomized to one of five groups:

1. Placebo daily for 7d after metronidazole treatment
2. LC-106 daily for 7d after metronidazole treatment
3. LC-106 daily for 3d + 4 days of placebo, starting after metronidazole treatment
4. LC-106 daily for 7d, starting on day 3 of metronidazole treatment
5. LC-115 daily for 7d after metronidazole treatment

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal individuals, 18- 40 years old
* BV by Amsel criteria (at least 3 of 4 criteria must be present)
* Abnormal Nugent score: ≥ 7
* Willing and able to provide written informed consent.
* HIV uninfected (by HIV Ab/Ag test at enrollment)
* Not pregnant by pregnancy test at enrollment, and unlikely to have an early pregnancy per clinician's assessment of last menstrual period and recent sexual activity.
* On continuous oral contraceptives (US site) or injectable progestin contraceptives (South African site) that suppress menstrual cycles, or willing to suppress menstrual cycles with one of these types of hormonal contraceptives
* Willing and able to attend study visits and comply with study procedures

Exclusion Criteria:

* History of clinically significant vaginal, cervical, or uterine disease including but not limited to: cancer of the female reproductive tract
* Prior hysterectomy
* Diagnosed with cervicovaginal infection (inclusive of gonorrhoeae, chlamydia, trichomonas) within the 30 days prior (or at enrollment visit). Yeast and bacterial vaginosis are not exclusionary.
* Use of antibiotics in the past 30 days
* Syphilis (positive screen at enrollment)
* Vulvovaginal candidiasis (positive microscopy at enrollment)
* Allergy to or contraindication to use of oral metronidazole
* High grade abnormal Pap (HSIL, AGC [Atypical Glandular Cells], ASCUS-H) at enrollment (LSIL, ASCUS, or HPV+ are all non-exclusionary)
* Currently participating in another study of an investigational product (excluding COVID vaccine studies)
* Use of long-acting systemic investigational product (e.g. injectable PrEP) within the past year
* Subject taking any of the following medications currently or in the past 30 days: systemic steroids (inhaled or nasal steroid therapy is permitted), interleukins, systemic interferons (e.g. local injection of interferon alpha for treatment of human papillomavirus is permitted) or systemic chemotherapy.
* History of coronary artery disease, myocardial infarction, chronic obstructive pulmonary disease, chronic renal failure, decompensated cirrhosis, or any other condition that in the opinion of the investigator will compromise ability to participate in the study.
* Use of an IUD (intrauterine device)
* Use of probiotics, prebiotics or synbiotics (supplements and products, oral or vaginal) within past 30 days. (NOTE: Oral yogurt with live cultures is allowed, as are fermented foods.)
* Active COVID-19 infection (determined by a positive PCR test of a nasal or nasopharyngeal swab) or recent exposure (< 14 days) to someone with confirmed COVID-19 infection (an exposure is considered being within 6 feet/180 cm of someone without a mask for more than 15 minutes). Potential participants who meet these criteria can delay screening until they have completed isolation or quarantine.
* Vaginal cleansing practices in the past 30 days (i.e. vaginal products for cleaning or drying, vaginal douching) (by eligibility questionnaire)
* Any other condition or situation that in the opinion of the investigator will compromise ability to participate in the study.
* Menopause: surgical; or absence of periods not due to hormonal contraception and in the setting of prior chemotherapy
* Use of testosterone for any reason
* Systolic blood pressure > 180 or diastolic blood pressure > 110 at screening or enrollment
* Hemoglobin < 9
* Less than 2 weeks since 2nd COVID vaccination (mRNA) or 1st vaccination (J&J) or booster
* Either breastfeeding/lactating or pregnant within 8 weeks prior to study entry

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-12-26 (Actual); Study Completion 2025-02-18 (Actual)

PRIMARY OUTCOMES:
Detection of LBP strains by metagenomic sequencing | Over 5 weeks
  Detection of any one strain from the LBP at 5% relative abundance or greater, or any combination of strains at 10% relative abundance or greater using shotgun metagenomic sequencing
Adverse events | Over 12 weeks
  Assessment of safety by comparing number and severity of adverse events

SECONDARY OUTCOMES:
Kinetics of colonization | Over 12 weeks
  Presence and quantity of each strain contained in the LBP measured by strain-specific quantitative PCR
Recurrent BV by Amsel and Nugent criteria | Over 12 weeks
  Presence of BV by Amsel criteria and/or Nugent criteria
Non-iners Lactobacillus dominance and abundance | Over 12 weeks
  Using 16S rRNA sequencing, relative abundance of non-iners Lactobacillus species in the vaginal fluid, and proportion with dominance by these species (> 50% relative abundance)
Alpha and beta diversity of the microbial community | Over 12 weeks
  Comparison of alpha and beta diversity metrics between arms before and after treatment with LBP
Proportion of participants reporting product was acceptable to use | Over 12 weeks
  Participant perceptions of and preferences for the vaginal LBP treatment

OTHER OUTCOMES:
Comparison of detection of LBP strains by metagenomics between US and South Africa | Over 12 weeks
  Comparison of all outcome measures at the US site vs. the South African site

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Mitchell, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (2):
- Massachusetts General Hospital, Boston, Massachusetts, United States
- CAPRISA - Vulindlela, Msunduzi Municipality, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data may be made available once primary and secondary analyses are completed, to investigators who request it.
Supporting Information: Study Protocol, SAP
Time Frame: Once primary and secondary analyses are completed.
Access Criteria: Requesters must have appropriate human subjects approval or waiver

REFERENCES:
- [Derived] Milford C, Dlamini BL, Mafunda NA, Hardwick TS, Lewis L, Khan AA, Mdladla MN, Mitchell CM, Potloane D. Bacterial Vaginosis [BV] knowledge, attitudes and behavioural changes after BV diagnosis among women enrolled in a clinical trial in Boston, USA and Vulindlela, South Africa: a qualitative study. BMC Womens Health. 2025 Dec 12;26(1):32. doi: 10.1186/s12905-025-04210-3. PMID 41382078
- [Derived] Chetty C, Mafunda N, Happel AU, Khan A, Cooley Demidkina B, Yende-Zuma N, Saidi Y, Mahabeer Polliah A, Lewis L, Osman F, Radebe P, Passmore JS, Kwon D, Ravel J, Ngcapu S, Liebenberg L, Symul L, Holmes S, Mitchell CM, Potloane D. Randomized trial of multi-strain Lactobacillus crispatus vaginal live biotherapeutic products after antibiotic therapy for bacterial vaginosis: study protocol for VIBRANT (vaginal lIve biotherapeutic RANdomized trial). Contemp Clin Trials Commun. 2025 Sep 16;48:101554. doi: 10.1016/j.conctc.2025.101554. eCollection 2025 Dec. PMID 41050878